CLINICAL TRIAL: NCT03651596
Title: Leveraging mHealth Messaging to Promote Adherence in Teens With CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00167162
Record Dates: First submitted 2018-08-24; First posted 2018-08-29 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Chronic Kidney Diseases; Adherence, Medication; Communication
Keywords: Adherence; Adolescence; mHealth
MeSH Terms: conditions — Renal Insufficiency, Chronic; Medication Adherence; Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard mHealth Messaging (Active Comparator): Individuals randomized to the Standard mHealth Messaging Group will receive a standard messaging intervention that has shown some efficacy in improving adherence in other samples.
  Interventions: Behavioral: Standard mHealth Messaging Group
- mHealth Messaging Intervention (Experimental): Individuals randomized to the mHealth Messaging Intervention Group will receive the newly developed messaging intervention.
  Interventions: Behavioral: mHealth Messaging Intervention Group

INTERVENTIONS:
Behavioral: mHealth Messaging Intervention Group — The newly developed intervention messages will be sent to individuals assigned to the intervention group during the study.
  Arms: mHealth Messaging Intervention
Behavioral: Standard mHealth Messaging Group — Standard mHealth messages will be sent to individuals assigned to the active control group during the study.
  Arms: Standard mHealth Messaging

SUMMARY:
The overall goal of this study is to develop and test effectively framed mobile health (mHealth) messages to promote medication adherence in teens with chronic kidney disease (CKD).

DETAILED DESCRIPTION:
Hypertension is a risk factor for chronic kidney disease (CKD) progression. Only 77% of adolescents with CKD are adherent to antihypertensive medications despite evidence that adherence slows disease progression. Mobile health (mHealth) applications show promise for improving adherence but most are not designed within health-promotion frameworks, only send medication reminders, use unreliable outcome measures, and/or have small effects on adherence. Nonadherence is a public health problem that may benefit from using health communication strategies to advance beyond reminders and improve mHealth efficacy. Highly effective health messages modify perceptions, attitudes, and skills to facilitate behavioral change; inappropriately framed messages (e.g., use of fear appeals) may have unintended, negative effects on health behaviors (i.e., reduce adherence). For adolescents with CKD, framing mHealth messages to motivate adherence may be a key factor in preventing disease progression; however, there has been little research to guide the use of this approach. Hence, the current study aims to develop and test effectively framed mobile health (mHealth) messages to promote medication adherence in teens with CKD.

Prior to study recruitment, the intervention messages will be developed by the research team and key stakeholders before testing in this pilot randomized controlled trial (RCT). Adolescents/young adults with CKD will be invited to participate in the pilot RCT to evaluate the intervention messages versus an active control condition; the primary outcome is antihypertensive medication adherence and secondary outcomes are participants' responses to surveys.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents/young adults aged 11-21 years
* Physician diagnosis of CKD stage 1-4
* Currently prescribed an antihypertensive medication and anticipate staying on an antihypertensive through the study duration (switching medication classes is permitted)
* Must have daily access to a Wi-Fi-enabled electronic device (e.g. iOS, Android 4.2 or higher, phone, tablet, computer) to receive private health information.

Exclusion Criteria:

* Adolescents/young adults who are on dialysis or had a kidney transplant
* Sibling participating in the study, unable to comprehend spoken English
* Cognitive delay precluding completion of study procedures
* And prescribed a liquid form of an antihypertensive medication (cannot be monitored).

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Antihypertensive medication adherence | 8 weeks during the study
  Electronic medication monitoring will be used to assess medication adherence, defined as the percentage of doses taken; higher percentages reflect that more doses were taken.

SECONDARY OUTCOMES:
Beliefs About Medication Scale | Up to 4 weeks before the study begins and up to 4 weeks after the study ends
  The construct, beliefs about medication, is measured with the Beliefs About Medication Scale. Mean scores are calculated for the the Positive Outcome Expectancies subscale (scale range = 1 to 7, higher scores indicate more positive beliefs) and the Negative Outcome Expectancies subscale (scale range = 1 to 7, higher scores indicate more negative beliefs).
Adolescent Medication Barriers Scale | Up to 4 weeks before the study begins and up to 4 weeks after the study ends
  The construct, barriers to adherence, is measured with the Adolescent Medication Barriers Scale (AMBS). The AMBS is reported as an overall mean score ranging from 1 to 5 with higher scores indicating more barriers to adherence.
Daily Medication Adherence Confidence Scale | Up to 4 weeks before the study begins and up to 4 weeks after the study ends
  The construct, medication adherence confidence, is measured with the Daily Medication Adherence Confidence Scale. This scale is reported as an overall mean score ranging from 1 to 10 with higher scores indicating more medication adherence confidence.
Daily Medication Adherence Importance and Motivation Scale | Up to 4 weeks before the study begins and up to 4 weeks after the study ends
  The construct, medication adherence importance and motivation, is measured with the Daily Medication Adherence Importance and Motivation Scale. The scale is reported as an overall mean score ranging from 1 to 10 with higher scores indicating higher daily medication adherence importance and motivation.
Self-reported Adherence | 8 weeks during the study
  Participants will be surveyed on whether the medication was taken or not (no=0, yes=1).
Impressions of Messages | 8 weeks during the study
  Participants will be surveyed on their impressions on the helpfulness of messages received (no=0, neither helpful nor unhelpful=1, yes=2).

CONTACTS AND LOCATIONS:
Overall Officials: Kristin A Riekert, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be shared in a de-identified form (i.e., clean, de-identified electronic database) upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon request.
Access Criteria: Data from this study will be shared in a de-identified form (i.e., clean, de-identified electronic database).

REFERENCES:
- [Derived] Eaton CK, Comer M, Pruette CS, Riekert KA. Medication adherence in youths with CKD: habits for success. Pediatr Nephrol. 2023 Nov;38(11):3791-3802. doi: 10.1007/s00467-023-05976-0. Epub 2023 Jun 12. PMID 37306720
- [Derived] Eaton C, Comer M, Pruette C, Psoter K, Riekert K. Text Messaging Adherence Intervention for Adolescents and Young Adults with Chronic Kidney Disease: Pilot Randomized Controlled Trial and Stakeholder Interviews. J Med Internet Res. 2020 Aug 14;22(8):e19861. doi: 10.2196/19861. PMID 32795983